CLINICAL TRIAL: NCT05117099
Title: Supplement: Long-term Effects of the Family Check-up on Depression and Suicide Across Trials and Development
Brief Title: Middle School Success Over Stress
Acronym: MSSOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3R01MH122213-01S1 (NIH)
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-01

CONDITIONS: Parenting; Parent-Child Relations; Depression; Self-regulation
MeSH Terms: conditions — Depression; Self-Control

STUDY DESIGN:
Intervention Model Description: Families will be assigned to treatment vs. waitlist control. The investigators will assess families at baseline and at 2-, 4-, and 6-month follow-ups. Families in the treatment condition will receive the intervention between baseline and the 2-month follow-up.The control group will receive the intervention following the 4-month assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCU Online + Coach (Experimental): Parents in this arm will receive access to the FCU Online website and telehealth coaching/ support provided by a trained mental health provider. The FCU Online website includes a brief 5-minute assessment, feedback on parents' responses, and online tools to support parenting in areas that were identified as challenges by the assessment. These tools include videos, animated videos, parenting tips, and interactives to help practice parenting skills.Telehealth coaching sessions will focus on Healthy Behaviors, Positive Parenting, Rules and Consequences, School Support, and Communication.
  Interventions: Behavioral: Family Check-Up
- Waitlist Control (No Intervention): Parents in this arm will initially serve as the control group but will receive access to the FCU Online website and telehealth coaching after completing three waves of data collection (baseline, 2-mo, and 4-mo follow-up).

INTERVENTIONS:
Behavioral: Family Check-Up — This intervention includes access to the Family Check-Up Online website and telehealth coaching provided by trained mental health providers. A minimum of 5 coaching sessions will be offered.
  Arms: FCU Online + Coach

SUMMARY:
It is clear that the COVID-19 pandemic has impacted families adversely in multiple ways, including economic stressors, mental health-related functioning, social/familial functioning, as well as responses to mandated safety measures (e.g. social distancing, stay-at-home orders, mask-wearing). Furthermore, families of school-age children have had to navigate online instruction and home schooling in the context of these difficult circumstances with little preparation for doing so effectively. School districts have varied widely in their ability to support parents during this crisis. These stressors are likely to have disproportionately adverse effects on lower-income and racial/ ethnic minority populations, for whom economic, academic, and family-level challenges were already pronounced. For instance, health effects of COVID-19 have hit African American and Latinx populations with disproportionate severity, including higher rates of hospitalization and death. Given the scale of pandemic impacts for families with school-aged children, the identification of effective family-focused interventions that target core mechanisms of change with a broad range of benefits for parents and youth across diverse populations, and that can be brought to scale rapidly and with fidelity, represent critical public health goals.

In this research study the investigators will adapt and test the efficacy of the Family Check-Up Online as a treatment to foster resilient family functioning in response to the COVID-19 pandemic. The investigators will test the effects of the adapted FCU Online program on key mechanisms of change that are predicted to directly impact child and family functioning: parenting skills, parental depression, and parent and child self-regulation. The investigators predict that changes in these key targets of the intervention will impact participant's response to the COVID-19 pandemic, including youth depression and behavior problems, the ability to cope with pandemic-focused stressors, and social/familial functioning.

ELIGIBILITY:
Inclusion Criteria:

* A caregiver must have a child between the ages of 10 and 14;
* the caregiver must be the parent or legal guardian of the participating youth;
* the caregiver must have a smartphone with text messaging capability and access to email; and
* the caregiver must score at least 1 or above on the Patient Health Questionnaire-2, or score at least 2 on any item of the Perceived Stress Scale-4.

Exclusion Criteria:

* the caregiver is unable to read in either English or Spanish;
* the child is unable to complete the survey without parent's help; or
* the family is already participating in another study of the University of Oregon's Prevention Science Institute.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stormshak, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon Prevention Science Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stormshak E, Connell A, Mauricio AM, McLaughlin M, Caruthers A. Digital Health Delivery of Parenting Skills to Improve Conduct Problems in Middle School Youth Across Two Distinct Randomized Trials. Prev Sci. 2025 May;26(4):582-591. doi: 10.1007/s11121-024-01750-2. Epub 2024 Nov 18. PMID 39556238
- [Derived] Mauricio AM, Hails KA, Caruthers AS, Connell AM, Stormshak EA. Family Check-Up Online: Effects of a Virtual Randomized Trial on Parent Stress, Parenting, and Child Outcomes in Early Adolescence. Prev Sci. 2024 Sep 24. doi: 10.1007/s11121-024-01725-3. Online ahead of print. PMID 39316242

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 377 families inquired about study participation. Some were excluded due to being unresponsive to outreach (n=191), declining to participate (n=11), or not meeting inclusion criteria (n=14). Families who returned baseline surveys (n=161 parent/caregivers; n=147 youth) were randomly assigned to one of two conditions.
Period: Baseline
Arm/Group | Waitlist Control | FCU Online + Coach
Started | 166 (87 parent participants and 79 youth participants) | 142 (74 parent participants and 68 youth participants)
Completed | 166 (87 parent participants and 79 youth participants) | 142 (74 parent participants and 68 youth participants)
Not Completed | 0 | 0
Period: 2-month Follow-up
Arm/Group | Waitlist Control | FCU Online + Coach
Started (Parent participants only.) | 73 | 70 (Parent participants only.)
Completed | 73 (Parent participants only.) | 70 (Parent participants only.)
Not Completed | 0 | 0
Period: 4-month Follow-up
Arm/Group | Waitlist Control | FCU Online + Coach
Started | 71 (Parent participants only.) | 63 (Parent participants only.)
Completed | 71 (Parent participants only.) | 63 (Parent participants only.)
Not Completed | 0 | 0
Period: 6-month Follow-up
Arm/Group | Waitlist Control | FCU Online + Coach
Started | 135 (73 parent participants and 62 youth participants) | 124 (69 parent participants and 55 youth participants)
Completed | 135 (73 parent participants and 62 youth participants) | 124 (69 parent participants and 55 youth participants)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: At baseline there were 87 families in the waitlist control condition and 74 in the FCU Online + Coach condition. Of the 87 families in the waitlist control condition, 87 parent/caregivers participated and 79 youth participated. Of the 74 families in the FCU Online + Coach condition, 74 parent/caregivers participated and 68 youth participated. Data entered in this section represent individuals, not dyads.
Groups:
- Total: Total of all reporting groups
Arm/Group | Waitlist Control | FCU Online + Coach | Total
Number analyzed (Participants) | 166 | 142 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: At baseline there were 87 families in the waitlist control condition and 74 in the FCU Online + Coach condition. Of the 87 families in the waitlist control condition, 87 parent/caregivers participated and 79 youth participated. Of the 74 families in the FCU Online + Coach condition, 74 parent/caregivers participated and 68 youth participated. Data entered in this section represent individuals, not dyads.
  years
    Parent: number analyzed (Participants) | 87 | 74 | 161
    Parent | 43.6 (7.09) | 41.91 (5.99) | 42.82 (6.64)
    Youth: number analyzed (Participants) | 79 | 68 | 147
    Youth | 12.44 (1.04) | 12.57 (1.06) | 12.50 (1.05)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Total participant population is comprised of parent and youth participants combined.
  Participants
    Parent: number analyzed (Participants) | 87 | 74 | 161
    Parent: Female | 82 | 70 | 152
    Parent: Male | 5 | 4 | 9
    Parent: Other | 0 | 0 | 0
    Parent: Prefer not to answer | 0 | 0 | 0
    Youth: number analyzed (Participants) | 79 | 68 | 147
    Youth: Female | 35 | 32 | 67
    Youth: Male | 34 | 34 | 68
    Youth: Other | 7 | 2 | 9
    Youth: Prefer not to answer | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: At baseline there were 87 families in the waitlist control condition and 74 in the FCU Online + Coach condition. Of the 87 families in the waitlist control condition, 87 parent/caregivers participated and 79 youth participated. Of the 74 families in the FCU Online + Coach condition, 74 parent/caregivers participated and 68 youth participated. Data entered in this section represent individuals, not dyads.
  Participants
    Parent: number analyzed (Participants) | 87 | 74 | 161
    Parent: Hispanic or Latino | 19 | 14 | 33
    Parent: Not Hispanic or Latino | 68 | 60 | 128
    Parent: Unknown or Not Reported | 0 | 0 | 0
    Youth: number analyzed (Participants) | 79 | 68 | 147
    Youth: Hispanic or Latino | 14 | 14 | 28
    Youth: Not Hispanic or Latino | 64 | 54 | 118
    Youth: Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: At baseline there were 87 families in the waitlist control condition and 74 in the FCU Online + Coach condition. Of the 87 families in the waitlist control condition, 87 parent/caregivers participated and 79 youth participated. Of the 74 families in the FCU Online + Coach condition, 74 parent/caregivers participated and 68 youth participated. Data entered in this section represent individuals, not dyads.
  Participants
    Parent: number analyzed (Participants) | 87 | 74 | 161
    Parent: American Indian or Alaska Native | 0 | 0 | 0
    Parent: Asian | 2 | 1 | 3
    Parent: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parent: Black or African American | 0 | 1 | 1
    Parent: White | 74 | 62 | 136
    Parent: More than one race | 9 | 10 | 19
    Parent: Unknown or Not Reported | 2 | 0 | 2
    Youth: number analyzed (Participants) | 79 | 68 | 147
    Youth: American Indian or Alaska Native | 1 | 0 | 1
    Youth: Asian | 4 | 1 | 5
    Youth: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Youth: Black or African American | 3 | 2 | 5
    Youth: White | 55 | 50 | 105
    Youth: More than one race | 9 | 13 | 22
    Youth: Unknown or Not Reported | 7 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 166 | 142 | 308

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Parent Mental Health and Well-being (Parent Report)
Description: Parents reported on their depressive symptoms using the Patient Health Questionnaire (PHQ-9), a 9-item brief depression screening questionnaire. Parents were asked to indicate the extent to which statements were true of their mood in the past two weeks using a 4-pt scale (not at all, several days, more than half the days, nearly every day). Scores ranged from 0-3. High scores indicate greater depressive symptoms.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: Number of participants differs between baseline and follow-up waves due to attrition (e.g., participants not returning follow-up surveys).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control | FCU Online + Coach
Number analyzed (Participants) | 87 | 74
score on a scale
  Baseline: number analyzed (Participants) | 86 | 74
  Baseline | .7442 (.53193) | .7523 (.61536)
  2-month Follow-up: number analyzed (Participants) | 73 | 70
  2-month Follow-up | .6484 (.50000) | .5571 (.51995)
  4-month Follow-up: number analyzed (Participants) | 71 | 63
  4-month Follow-up | .6182 (.42444) | .4903 (.54089)
  6-month Follow-up: number analyzed (Participants) | 72 | 68
  6-month Follow-up | .5386 (.46832) | .5359 (.61996)
Statistical Analysis 1: Comparison: Waitlist Control vs FCU Online + Coach; Test type: Superiority; p = .548, ANOVA

2. Primary Outcome: Change From Baseline in Parental Stress (Parent Report)
Description: Parents reported on their parenting stress using the Parenting Stress Index (PSI), a 14-item questionnaire. Parents were asked to indicate the extent to which statements were true of their experience in the past month using a 5-pt scale (never, almost never, sometimes, fairly often, very often). Scores ranged from 0-4. High scores indicate greater parenting stress.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control | FCU Online + Coach
Number analyzed (Participants) | 86 | 73
score on a scale
  Baseline | 1.8205 (.50818) | 1.8341 (.61821)
  2-month Follow-up: number analyzed (Participants) | 73 | 70
  2-month Follow-up | 1.8033 (.51930) | 1.5365 (.60099)
  4-month Follow-up: number analyzed (Participants) | 71 | 63
  4-month Follow-up | 1.7616 (.50651) | 1.5351 (.64845)
  6-month Follow-up: number analyzed (Participants) | 72 | 68
  6-month Follow-up | 1.6619 (.46722) | 1.5575 (.67258)

3. Primary Outcome: Change From Baseline in Child Behavior and Emotional Problems (Parent Report)
Description: Parents reported on their child's problem behavior using the Strengths and Difficulties Questionnaire (SDQ), a 25-item brief behavioral screening questionnaire that consists of 5 subscales with 5 questions each. The 5 subscales are conduct problems, emotional problems, hyperactivity, peer problems, and prosocial behavior. Parents were asked to indicate the extent to which statements were true of their child's behavior in the past month using a 3-pt scale (not true, somewhat true, and certainly true). Response options for each item ranged from 0-2. Subscale totals were created by summing responses for a possible range of 0-10 for each subscale. The sums from each subscale were summed to create a composite score. High scores indicate greater conduct problems.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control | FCU Online + Coach
Number analyzed (Participants) | 87 | 74
score on a scale
  Baseline | 13.2184 (6.48330) | 14.2568 (7.53814)
  2-month Follow-up: number analyzed (Participants) | 73 | 70
  2-month Follow-up | 12.8630 (6.62343) | 12.2143 (6.32660)
  4-month Follow-up: number analyzed (Participants) | 71 | 63
  4-month Follow-up | 11.6056 (6.23465) | 12.1587 (7.17119)
  6-month Follow-up: number analyzed (Participants) | 73 | 69
  6-month Follow-up | 11.9726 (5.93243) | 12.2319 (7.50910)
Statistical Analysis 1: Comparison: Waitlist Control vs FCU Online + Coach; Test type: Superiority; p = .915, ANOVA

4. Primary Outcome: Change From Baseline in Youth Depression (Parent Report)
Description: Parents reported on their child's depressive symptoms using the Patient Health Questionnaire (PHQ-9), a 9-item brief depression screening questionnaire. Parents were asked to indicate the extent to which statements were true of their child's mood in the past two weeks using a 4-pt scale (not at all, several days, more than half the days, nearly every day). Scores ranged from 0-3. High scores indicate greater depressive symptoms.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control | FCU Online + Coach
Number analyzed (Participants) | 87 | 74
score on a scale
  Baseline | .6092 (.54218) | .6937 (.59356)
  2-month Follow-up: number analyzed (Participants) | 73 | 70
  2-month Follow-up | .5219 (.49215) | .5423 (.51117)
  4-month Follow-up: number analyzed (Participants) | 71 | 63
  4-month Follow-up | .4589 (.46516) | .4925 (.51814)
  6-month Follow-up: number analyzed (Participants) | 73 | 69
  6-month Follow-up | .4810 (.47972) | .4783 (.51213)
Statistical Analysis 1: Comparison: Waitlist Control vs FCU Online + Coach; Test type: Superiority; p = .663, ANOVA

5. Primary Outcome: Change From Baseline in Parenting Skills (Parent Report)
Description: Parents reported on their parenting skills using a version of the Parenting Young Children Questionnaire (PARYC). The PARYC version adapted for this study was a 21-item questionnaire. Parents were asked to indicate the extent to which statements were true of their child's behavior in the past month using a 5-pt scale (never, rarely, sometimes, often, and very often). Scores for each item ranged from 0-4, and scores were averaged to create a total score. High scores indicate greater parenting skills.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control | FCU Online + Coach
Number analyzed (Participants) | 87 | 74
score on a scale
  Baseline | 2.9253 (.66703) | 2.9122 (.72319)
  2-month Follow-up: number analyzed (Participants) | 72 | 70
  2-month Follow-up | 2.8611 (.74693) | 3.1286 (.65212)
  4-month Follow-up: number analyzed (Participants) | 71 | 62
  4-month Follow-up | 2.9155 (.71707) | 3.1532 (.64394)
  6-month Follow-up: number analyzed (Participants) | 72 | 67
  6-month Follow-up | 2.9375 (.74085) | 2.9627 (.69257)
Statistical Analysis 1: Comparison: Waitlist Control vs FCU Online + Coach; Test type: Superiority; p = .138, ANOVA

6. Primary Outcome: Change From Baseline in Positive Family Relationships (Parent Report)
Description: Parents reported on their family relationships using a "family togetherness" scale adapted from the Community Action for Successful Youth (CASEY) questionnaire. The scale used for this study consisted of 3 items. Parents were asked to indicate the extent to which statements were true of their experience in the past month using a 5-pt scale (never true, sometimes true, true about half the time, often true, and always true). Scores ranged from 1-5. High scores indicate greater positive family relationships.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control | FCU Online + Coach
Number analyzed (Participants) | 86 | 74
score on a scale
  Baseline | 3.3798 (.85888) | 3.4189 (.88804)
  2-month Follow-up: number analyzed (Participants) | 73 | 70
  2-month Follow-up | 3.3014 (.80539) | 3.6833 (.91161)
  4-month Follow-up: number analyzed (Participants) | 71 | 63
  4-month Follow-up | 3.4437 (.72097) | 3.7566 (.94888)
  6-month Follow-up: number analyzed (Participants) | 73 | 68
  6-month Follow-up | 3.5662 (.82904) | 3.5637 (.97609)
Statistical Analysis 1: Comparison: Waitlist Control vs FCU Online + Coach; Test type: Superiority; p = .114, ANOVA

7. Primary Outcome: Change From Baseline in Family Conflict (Parent Report)
Description: Parents reported on their family conflict using a "family conflict" scale adapted from the Community Action for Successful Youth (CASEY) questionnaire. The scale used for this study consisted of 4 items. Parents were asked to indicate the extent to which statements were true of their experience in the past month using a 7-pt scale (never, once, twice, 3 times, 4 or 5 times, 6 or 7 times and more than 7 times). Scores for each item ranged from 0-6, and scores were averaged to create a total score. High scores indicate increased family conflict.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control | FCU Online + Coach
Number analyzed (Participants) | 87 | 74
score on a scale
  Baseline | 1.8046 (1.14908) | 1.8559 (1.01044)
  2-month Follow-up: number analyzed (Participants) | 73 | 70
  2-month Follow-up | 1.7637 (1.13414) | 1.5202 (.95062)
  4-month Follow-up: number analyzed (Participants) | 71 | 63
  4-month Follow-up | 1.6725 (.96602) | 1.3254 (.97202)
  6-month Foll1.4338ow-up: number analyzed (Participants) | 73 | 68
  6-month Foll1.4338ow-up | 1.5696 (1.03040) | 1.4338 (1.10934)
Statistical Analysis 1: Comparison: Waitlist Control vs FCU Online + Coach; Test type: Superiority; p = .065, ANOVA

8. Primary Outcome: Change From Baseline in Youth Depression (Child Report)
Description: Youth reported on their depressive symptoms using the Patient Health Questionnaire (PHQ-9), a 9-item brief depression screening questionnaire modified for teen use. Youth were asked to indicate the extent to which statements were true of their mood in the past two weeks using a 4-pt scale (not at all, several days, more than half the days, nearly every day). Scores for each item ranged from 1-4, and scores were averaged to create a total score. High scores indicate greater depressive symptoms.
Time Frame: baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control | FCU Online + Coach
Number analyzed (Participants) | 79 | 68
score on a scale
  Baseline | 1.7708 (.71537) | 1.6029 (.62672)
  6-month Follow-up: number analyzed (Participants) | 61 | 55
  6-month Follow-up | 1.8070 (.73077) | 1.7596 (.69644)
Statistical Analysis 1: Comparison: Waitlist Control vs FCU Online + Coach; Test type: Superiority; p = .394, ANOVA

9. Primary Outcome: Change From Baseline in Positive Family Relationships (Child Report)
Description: Youth reported on their family relationships using a "family togetherness" scale adapted from the Community Action for Successful Youth (CASEY) questionnaire. The scale used for this study consisted of 3 items. Youth were asked to indicate the extent to which statements were true of their experience in the past month using a 5-pt scale (never true, sometimes true, true about half the time, often true, and always true). Scores ranged from 1-5. High scores indicate greater positive family relationships.
Time Frame: baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control | FCU Online + Coach
Number analyzed (Participants) | 77 | 67
score on a scale
  Baseline | 3.6061 (1.06613) | 3.5699 (1.10865)
  6-month Follow-up: number analyzed (Participants) | 62 | 55
  6-month Follow-up | 3.4453 (1.15739) | 3.4909 (1.17563)
Statistical Analysis 1: Comparison: Waitlist Control vs FCU Online + Coach; Test type: Superiority; p = .388, ANOVA

10. Primary Outcome: Change From Baseline in Family Conflict (Child Report)
Description: Youth reported on their family conflict using a "family conflict" scale adapted from the Community Action for Successful Youth (CASEY) questionnaire. The scale used for this study consisted of 4 items. Youth were asked to indicate the extent to which statements were true of their experience in the past month using a 7-pt scale (never, once, twice, 3 times, 4 or 5 times, 6 or 7 times and more than 7 times). Scores ranged from 1-7. High scores indicate increased family conflict.
Time Frame: baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control | FCU Online + Coach
Number analyzed (Participants) | 76 | 68
score on a scale
  Baseline | 2.6184 (1.22234) | 2.8640 (1.31043)
  6-month Follow-up: number analyzed (Participants) | 62 | 55
  6-month Follow-up | 2.5323 (1.13394) | 2.6636 (1.08463)
Statistical Analysis 1: Comparison: Waitlist Control vs FCU Online + Coach; Test type: Superiority; p = .332, ANOVA

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events over the study period (until their 6-month post-test was completed).
Groups:
- Waitlist Control- Parents: Includes parents randomized to waitlist control.
- FCU Online + Coach- Parents: Includes parents randomized to FCU Online + Coaching.
- Waitlist Control- Youth: Includes youth randomized to waitlist control.
- FCU Online + Coach- Youth: Includes youth randomized to FCU Online + Coaching.
Arm/Group | Waitlist Control- Parents | FCU Online + Coach- Parents | Waitlist Control- Youth | FCU Online + Coach- Youth
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/74 | 0/79 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/74 | 0/79 | 0/68
Other Adverse Events (participants affected / at risk) | 0/87 | 0/74 | 0/79 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT05117099/Prot_SAP_002.pdf
  • Informed Consent Form (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT05117099/ICF_001.pdf